CLINICAL TRIAL: NCT04318730
Title: Phase II Study for Combination of Camrelizumab and Apatinib in the Second-line Treatment of Recurrent or Metastatic Adrenocortical Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Associate Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR1900028111
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Adrenocortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab was administered 200mg iv every 3 weeks, Apatinib was administered 250 mg p.o. qd.
  Other Names: Apatinib

SUMMARY:
Adrenocortical carcinoma (ACC) is a rare aggressive malignant tumor. According to the literature, the 5-year survival rate of ACC is 12%-47%. For patients with advanced ACC, mitotane alone or combined with traditional chemotherapy was the first-line standard treatment, but its progression-free survival was only about 1 year. However, for patients who fail the first-line treatment, there is a lack of effective treatment. For ACC patients who had failed first-line chemotherapy, a phase II clinical trial found that the objective response rate and the disease control rate of PD-1 inhibitor Keytruda were 14% and 64% respectively, and no grade 3 or 4 adverse events were observed. Anti-tumor angiogenic drugs combined with PD-1 inhibitors have shown impressive clinical data in many solid tumors. This study is aimed to evaluate the efficacy and safety of PD-1 inhibitor camrelizumab combined with apatinib in patients with recurrent or metastatic ACC after standard treatment failure, and to seek new treatment for this population.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of adrenocortical carcinoma;
2. Patients with metastatic or inoperable adrenocortical carcinoma that has progressed, metastasized, or recurred after first-line standard treatment (mitotane monotherapy, chemotherapy alone, mitotane combined chemotherapy);
3. Aged >=18 years;
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
5. At least one measurable lesion, according to RECIST 1.1;
6. Major organ functions within 28 days prior to treatment meet the following criteria(14 days without transfusion): HB≥80g/L, ANC≥1.5x10^9/L, PLT ≥80x10^9/L; TBIL≤1.5 ULN, ALT and AST ≤2.5 ULN, if there exists hepatic metastases, ALT and AST ≤5 ULN, Cr ≤1.5 ULN or CCr ≥60ml/min; INR or PT ≤1.5 ULN, APTT ≤1.5 ULN (if the patient is receiving anticoagulant therapy, PT and APTT should be within the expected treatment range); Cardiac Markers and BNP≤ULN；TSH≤ULN (If TSH is abnormal, T3 and T4 should be normal)
7. Appropriate contraception should be used from the start of treatment to 120 days after the end of treatment;
8. Have signed consent form.

Exclusion Criteria:

1. Patients with another primary malignancy within 5 years prior to starting the study drug, except for cured in situ cervical carcinoma and cured non-melanoma skin cancer;
2. Have central nervous system metastasis with symptoms and need hormonal intervention;
3. Had received strong CYP3A4 inhibitors within one week prior to enrollment or received strong CYP3A4 inducers within two weeks prior to enrollment;
4. Poor control of high blood pressure (SBP>140mmHg or DBP>90mmHg);
5. Congestive heart failure of New York Heart Association (NYHA) Class III or IV;
6. Thromboembolic events occurred within 1 year prior to enrollment;
7. ECG QT interval >500ms;
8. Previous systemic immunosuppressive therapy;
9. Previous anti-PD-1, anti-PD-L1 antibody or anti- CTLA-4 antibody treatment;
10. Received TKI treatment within 2 weeks prior to starting the study drug;
11. Participate in clinical trials of other interventional drugs within 4 weeks prior to starting the study drug;
12. Received systemic therapy with corticosteroids or other immunosuppressants within 2 weeks prior to starting the study drug;
13. An anti-tumor vaccine or a live vaccine was given within 4 weeks prior to starting the study drug;
14. Major surgery or severe trauma within 4 weeks prior to starting the study drug;
15. Severe infections occurred within 4 weeks prior to starting the study drug;
16. Have an active autoimmune disease or a history of autoimmune diseases;
17. Have a history of immunodeficiency;
18. Have an active tuberculosis infection;
19. Have active hepatitis;
20. Patients with symptoms of gastrointestinal bleeding or risk of bleeding;
21. Active infection, or patients are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | up to 60 months
  The rate of complete response and partial response.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhu YC, Wei ZG, Wang JJ, Pei YY, Jin J, Li D, Li ZH, Liu ZR, Min Y, Li RD, Yang L, Liu JY, Wei Q, Peng XC. Camrelizumab plus apatinib for previously treated advanced adrenocortical carcinoma: a single-arm phase 2 trial. Nat Commun. 2024 Nov 29;15(1):10371. doi: 10.1038/s41467-024-54661-9. PMID 39609453